CLINICAL TRIAL: NCT07067541
Title: Clinical Observation of Topical Lidocaine Cream Combined With Moisturizing Cream in the Treatment of Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Tang Junting, Director, First Affiliated Hospital of Kunming Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-L-88
Record Dates: First submitted 2025-07-01; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Drug: Control lidocaine cream
- Experimental group (Experimental)
  Interventions: Drug: Experimental lidocaine cream + moisturizer cream

INTERVENTIONS:
Drug: Control lidocaine cream — lidocaine cream alone
  Arms: Control Group
Drug: Experimental lidocaine cream + moisturizer cream — lidocaine cream + moisturizer cream
  Arms: Experimental group

SUMMARY:
Twenty-five patients with atopic dermatitis applied lidocaine cream plus a moisturizer to the right limb and lidocaine cream alone to the left limb, twice daily for four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-65 years.
2. Clinical diagnosis of atopic dermatitis according to the 2020 Guidelines for the Diagnosis and Treatment of Atopic Dermatitis in China (symmetrical eczematous lesions for ≥6 months plus personal/family atopy history or elevated IgE/eosinophilia).
3. Voluntarily signed informed consent form.

Exclusion Criteria:

1. Active heart, liver, kidney, or other serious systemic illness.
2. History of viral or bacterial infection within 1 month prior to enrollment.
3. Immunocompromised patients or those receiving systemic immunosuppressive therapy.
4. Known allergy to lidocaine, moisturizer components, or any study-related topical agents.
5. Pregnant or breastfeeding women.
6. Use of topical corticosteroids or calcineurin inhibitors within 2 weeks prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
change in SCORAD (SCORing Atopic Dermatitis) from baseline | 4 weeks
  For each patient, a score will be obtained at baseline, after 4 weeks. The minimum score is 0 (best outcome) and the maximum score is 103 (worst outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China